CLINICAL TRIAL: NCT01045200
Title: Nurse-or Surgeon-led Follow-up After Rectal Cancer: a Randomised Trial.
Brief Title: Nurse-or Surgeon-led Follow-up After Rectal Cancer
Status: Completed | Type: Observational
Sponsor: Centrallasarettet Västerås (Other)
Responsible Party: Kenneth Smedh MD, PhD, Head of Colorectal Surgery, Department of Surgery, Central Hospital, Västerås, Sweden
Other Study IDs: DNR 01-498
Record Dates: First submitted 2010-01-06; First posted 2010-01-08 (Estimated); Last update posted 2010-01-08 (Estimated); Status verified 2002-01

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; follow-up; specialist nurse
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Follow-up: Patients curatively operated for rectal cancer
  Interventions: Other: Comparison of follow-up

INTERVENTIONS:
Other: Comparison of follow-up — Comparison of follow-up by nurse or surgeon after rectal cancer surgery
  Other Names: Rectal cancer patients

SUMMARY:
Follow-up programmes consume a large amount of resources with less time for the surgeon to take on new patients. The aim of this randomised study was to compare patient satisfaction, resource utilisation, and medical safety in patients curatively operated for rectal cancer that were followed-up by a surgeon or a nurse.

ELIGIBILITY:
Inclusion Criteria:

* Patients curatively operated for rectal cancer.
* Patients had to be more than 18 years of age and written and oral informed consent was obtained.

Exclusion Criteria:

* Those with psychiatric disorders, dementia and whose general condition had deteriorated with an expected survival of less than six months were not eligible.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Operated for rectal cancer at the colorectal unit of the Central Hospital in Västerås, Sweden.
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2002-01; Primary Completion 2004-10 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | At each patient visit, i.e. every 6 months during the first three years than every year after rectal cancer surgery.

SECONDARY OUTCOMES:
Resource utilisation | at each patient visit, i.e. every 6 months during the first three years than every year after rectal cancer surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Departement of Surgery, Central Hospital, Västerås, Sweden